CLINICAL TRIAL: NCT07283341
Title: The Role of Diet and Gastrointestinal Motility in Irritable Bowel Syndrome (IBS)
Brief Title: Diet and Motility in IBS
Acronym: IBS
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 22-020433
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Irritable Bowel Syndrome (IBS)
Keywords: Irritable Bowel Syndrome; Diet; Motility; Wireless Patch System
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IBS Cohort: Participants ages 8 to 18 years old who meet Rome IV diagnostic criteria for IBS
  Interventions: Diagnostic Test: Wireless Patch System
- Control Cohort: Participants ageds 8-18 years old who don't have IBS
  Interventions: Diagnostic Test: Wireless Patch System

INTERVENTIONS:
Diagnostic Test: Wireless Patch System — The Wireless Patch System will be placed on the abdominal skin. Participants will receive an iPhone containing the WPS app to record symptoms and meals. Participants undergoing a clinically indicated dietary intervention will complete study procedures before and after the dietary intervention.

SUMMARY:
The goal of this observational study is to identify factors that influence symptoms in children with irritable bowel syndrome (IBS), to find ways to make diet treatments work better and possibly create personalized plans to help each child with IBS feel better. The main question it aims to answer is:

1. What types of food do the kids eat and how do these diets relate to their symptoms?
2. Is there any motility pattern that we can identify from the kids with or without IBS using a wearable patch?
3. What kinds of bacteria and chemicals are found in the gut and urine of children with IBS, and how are these linked to their IBS symptoms?

Participants will use the wearable patch, answer questionnaires, collect stool and urine samples, and recall their 24 hours dietary.

ELIGIBILITY:
Inclusion Criteria:

Cases:

1. Males and females age 8 - 18 years
2. Diagnosis of irritable bowel syndrome (IBS).
3. Parental/guardian permission (informed consent) and child assent

Controls:

1. Males and Females age 8-18 years
2. No diagnosis of abdominal pain disorder
3. Parental/guardian permission (informed consent) and child assent

Exclusion Criteria:

Cases:

1. Allergy to adhesives
2. Inability to cooperate with study design
3. Antibiotic intake in the past 4 weeks
4. Inflammatory gastrointestinal disorder diagnosis

Controls:

1. Allergy to adhesives
2. Inability to cooperate with study design
3. Antibiotic intake in the past 4 weeks
4. Inflammatory gastrointestinal disorder diagnosis

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants meet the eligibility criteria listed.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Gut myoelectric activity in children with IBS and controls using the non-invasive wireless patch system (WPS) | Approximately one year.
  Differences in total activity, pre- and post-prandial activity ratios, nighttime colonic activity, and night-to-day colonic activity ratios between IBS patients and controls. WPS reading will be completed after each study visit. Differences will be compared at the 3rd and 4th quarters of each year.

CONTACTS AND LOCATIONS:
Overall Officials: Alain Benitez, MD, MSTR, Principal Investigator — Children's Hospital of Philadelphia, University of Pennsylvania
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Axelrod L, Axelrod S, Navalgund A, Triadafilopoulos G. Pilot Validation of a New Wireless Patch System as an Ambulatory, Noninvasive Tool That Measures Gut Myoelectrical Signals: Physiologic and Disease Correlations. Dig Dis Sci. 2021 Oct;66(10):3505-3515. doi: 10.1007/s10620-020-06663-y. Epub 2020 Oct 15. PMID 33063188